CLINICAL TRIAL: NCT03198416
Title: Assessment Of Pharyngeal Anatomy In Obstructive Sleep Apnea With High Resolution Manometry
Brief Title: Pharyngeal Anatomy In Obstructive Sleep Apnea With HRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, David Kent, Assistant Professor, Department of Otolaryngology, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 170755
Record Dates: First submitted 2017-06-11; First posted 2017-06-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: All patients who meet eligiblity will undergo HRM at the same time as the operative DISE procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Investigational Device (Experimental): Consented participants who meet eligibility will have a drug induced sleep endoscopy (DISE) with the Solar GI High Resolution pharyngeal Manometry system.
  Interventions: Device: High-resolution pharyngeal manometry catheter

INTERVENTIONS:
Device: High-resolution pharyngeal manometry catheter — The system is a widely-used tool in gastrointestinal medicine for high resolution mapping of pressures within tubular organs.The device will be deployed trans-nasally into the pharyngeal and esophageal lumen in exactly the same fashion as is done for motility studies.

SUMMARY:
This is a single-arm study involving the use of a high resolution manometry (HRM) diagnostic device that is not utilized in any clinical decision-making processes. All patients scheduled for DISE as part of their regular clinical care will be screened for enrollment via described inclusion and exclusion criteria.

DETAILED DESCRIPTION:
High-resolution pharyngeal manometry (HRM) is a diagnostic technique that has the potential to objectively measure pharyngeal collapse patterns in obstructive sleep apnea (OSA) during sedation as well as natural sleep. The purpose of this study is to assess the utility of HRM in objectively mapping patterns of pharyngeal collapse observed during drug-induced sleep endoscopy (DISE). Quantifying pharyngeal collapse patterns that occur during sedation and in natural sleep may significantly impact the selection and success of surgical treatments, as well as surgical outcome assessment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years old)
* A diagnosis of obstructive sleep apnea as determined by polysomnogram with an apnea-hypopnea index of ≥ 5.0/hr
* Intolerant of continuous positive airway pressure (CPAP) therapy due to physical or psychosocial limitations as determined by PI
* Scheduled to undergo DISE as part of routine clinical assessment for further evaluation of pharyngeal anatomy

Exclusion Criteria:

* Patient is unable to consent for research due to a pre-existing neurologic condition as determined by PI
* Patient is unable to consent for research due to language barriers
* Patient has a history of egg allergy as determined by history or self- report
* Patient is pregnant as determined by patient report or preoperative anesthesia evaluation
* Cardiopulmonary or other medical conditions precluding safe sedation as determined by clinical history and exam
* History of palatal or pharyngeal airway surgery except tonsillectomy as determined by clinical history and exam
* History of radiation treatment to the head or neck as determined by clinical history and/or exam
* Severe nasal airway obstruction preventing simultaneous flexible nasopharyngoscopy and manometry probe insertion as determined by physical exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Pharyngeal pressure differentials | Collected during operative procedure, taking about 15 minutes.
  A high-resolution pharyngeal manometry catheter will be used to capture air pressure data in millimeters of mercury at 0.8mm intervals throughout the pharynx and proximal esophagus during the drug-induced sleep endoscopy procedure. This data will be used to generate maps of pressure data over time.
Video endoscopy of pharyngeal collapse | Collected during operative procedure, the video endoscopy will take about 15 minutes.
  Video from the flexible nasopharyngoscopy exam conducted during the drug-induced sleep endoscopy will be recorded and time-synched to the high-resolution pharyngeal manometry catheter output. The video results will be graded by a trained reviewer using a validated scoring system called the VOTE classification. The VOTE system is a subjective scoring system based on video endoscopy that scores the degree and configuration of airway obstruction related to the velum (soft palate), oropharyngeal lateral walls, tongue base, and epiglottis. The VOTE classification results will be compared to the pressure catheter results to examine for correlations.

SECONDARY OUTCOMES:
Patient tolerance of catheter | Completed pre-operatively, after catheter insertion, taking less than 5 minutes.
  Patient comfort as indicated by pre operative pain survey
Patient tolerance of catheter | Completed at follow up visit about 1 week post-operative, taking less than 5 minutes.
  Patient comfort as indicated by post operative pain survey

CONTACTS AND LOCATIONS:
Overall Officials: David T. Kent, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kent DT, Scott WC, Ye C, Fabbri D. Objective Pharyngeal Phenotyping in Obstructive Sleep Apnea With High-Resolution Manometry. Otolaryngol Head Neck Surg. 2023 Jul;169(1):164-175. doi: 10.1002/ohn.257. Epub 2023 Jan 29. PMID 36939475